CLINICAL TRIAL: NCT05628675
Title: Feasibility of a Psychoeducational Group Intervention to Improve Parental Reflective Functioning and Bonding in Prenatal Depression
Brief Title: A Prenatal Bonding Intervention for Pregnant Women With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R&D2022/056; 302132 (Other: IRAS)
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2022-08

CONDITIONS: Depression; Pregnancy
Keywords: Prenatal Bonding; Reflective Functioning; Maternal-Foetal Attachment; Mentalisation; Prenatal Depression; Perinatal Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Single-arm repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single-session 90-minute psychoeducational group ("Baby CHAT") delivered antenatally.
  Interventions: Other: Baby CHAT

INTERVENTIONS:
Other: Baby CHAT — Baby CHAT is an approximately 90-minute group intervention to be delivered during pregnancy. The group is comprised of psychoeducational material about a baby's social development after birth and while the baby is growing in the womb. Attendees are encouraged to think about when an infant's social development begins and consider whether this occurs before or after birth. Participants are then shown a video clip of Reissland et al.'s (2016) study showing 4D ultrasound images of foetuses mouthing in response to sounds that are presented to them outside the womb. During Baby CHAT, parents are encouraged to reflect on this information in the context of their own baby's development, including their likes and dislikes, routine and personality. The final section of the group involves generating ideas for social activities that parents can try with their baby prior to birth, such as singing to, massaging or reading to their baby.

SUMMARY:
The goal of this clinical trial is to test a group for pregnant women with depression that aims to help them build a stronger relationship with their unborn baby. The main questions it aims to answer are:

* Is the group acceptable to pregnant women with depression?
* Is it possible to run this group with pregnant women with depression?
* Could the group potentially impact bonding, parental reflective functioning and mood?

Participants will be asked to:

* attend the group (which lasts 90mins)
* complete questionnaires before and after the group, and 1 month later

DETAILED DESCRIPTION:
Depression during pregnancy is a common mental health problem. Pregnant women with depression often continue to feel depressed after their baby is born, which can have several negative effects for both mother and child. For example, depressed mothers can find it harder to build a good relationship with their baby. Existing treatments for depression may not be sufficient to also improve the relationship between mother and baby. Depressed mothers may therefore need more specific help with connecting to their baby.

One promising new intervention is Baby CHAT. Baby CHAT is a single-session group that helps expectant parents learn about their unborn baby by viewing moving 4D ultrasound scans. It is believed that this will help parents to build a stronger relationship with their unborn baby. Baby CHAT has already been trialled with parents without any mental health problems, with promising results. This study aims to assess whether Baby CHAT is helpful for pregnant women with depression, collect data to inform future large-scale trials, and to develop the intervention from participants' feedback. The main research question asks: is Baby CHAT acceptable and feasible to deliver with pregnant women with depression?

Participants eligible to take part in the project will be people aged ≥18 years who are pregnant, between 20- and 34-weeks' gestation, and currently experiencing depressive symptoms. The project is taking place at an NHS site, with participants recruited from mental health and maternity services and online advertising. Participants will attend an online Baby CHAT group and complete online questionnaires at three time points (before and after Baby CHAT, and at one-month follow-up). The questionnaires will assess participants' relationship with their unborn baby, their ability to imagine their unborn baby as a separate person, and their level of depressive symptoms. The anticipated study end date is May 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Currently pregnant
2. Aged ≥18 years
3. Between 20- and 34-weeks' gestation
4. Currently experiencing depressive symptoms as identified by the Edinburgh Postnatal Depression Scale (EPDS)
5. Resident in or accessing services in a London borough served by South London & Maudsley NHS Foundation Trust

Exclusion Criteria:

1. Experiencing severe depression or current severe co-morbid diagnoses e.g. psychosis
2. Endorse 'yes, quite often' or 'sometimes' on question 10 of the Edinburgh Postnatal Depression Scale (EPDS; in the past 7 days, 'the thought of harming myself has occurred to me') at screening
3. Unable to complete informed consent and the questionnaires in English

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Cockburn, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 21
Completed | 18
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Asian British | 1
  Black or Black British | 3
  Mixed ethnic group | 1
  White or White British | 13
  Other ethnic group | 2
Gestational age at baseline [Mean (Standard Deviation); unit: weeks] | 29.1 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change on Maternal Antenatal Attachment Scale (MAAS)
Description: The Maternal Antenatal Attachment Scale (MAAS; Condon, 1993) is a self-report questionnaire for expectant mothers, designed to assess the maternal-foetal attachment during pregnancy. The scale consists of 19 items on a 5-point Likert scale assessing women's attitudes, feelings and behaviours towards their foetus. Higher total scores indicate stronger prenatal bonding i.e. a better outcome (range 19-95).
Time Frame: Baseline, up to 48-hours post-intervention, 1-month follow-up
Population: N=4 delivered their babies by Time 3 and therefore did not complete the MAAS at this timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
score on a scale
  Time 1 (pre-intervention) | 69.7 (9.1)
  Time 2 (up to 48-hours post-intervention) | 72.4 (7.9)
  Time 3 (1-month follow-up): number analyzed (Participants) | 15
  Time 3 (1-month follow-up) | 75.9 (8.0)
Statistical Analysis 1: Comparison: Intervention; Effect size calculation from Time 1 to Time 2 on MAAS; Test type: Other; Effect size (Hedge's g) = 0.32, 95% CI 2-sided [-0.33 to 0.96]
Statistical Analysis 2: Comparison: Intervention; Effect size calculation from Time 1 to Time 3 on MAAS; Test type: Other; Effect size (Hedge's g) = 0.72, 95% CI 2-sided [0.02 to 1.42]

2. Secondary Outcome: Change on Prenatal Parental Reflective Functioning Questionnaire (P-PRFQ)
Description: The Prenatal Parental Reflective Functioning Questionnaire (P-PRFQ; Pajulo et al., 2015) is a 14-item self-report questionnaire assessing expectant parents' abilities to think of their foetus as a separate individual with a developing temperament, personality and needs. The scale can be used during the second and third trimester of pregnancy. Higher total scores indicate stronger prenatal parental reflective functioning i.e. a better outcome (range 14-98).
Time Frame: Baseline, up to 48-hours post-intervention, 1-month follow-up
Population: N=1 delivered their baby before fully completing Time 2 and a total N=4 had delivered their babies by Time 3, therefore not completing the P-PRFQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
score on a scale
  Time 1 (pre-intervention) | 60.7 (15.1)
  Time 2 (up to 48-hours post-intervention): number analyzed (Participants) | 18
  Time 2 (up to 48-hours post-intervention) | 65.7 (11.7)
  Time 3 (1-month follow-up): number analyzed (Participants) | 15
  Time 3 (1-month follow-up) | 67.1 (10.1)
Statistical Analysis 1: Comparison: Intervention; Effect size calculation from Time 1 to Time 2 on P-PRFQ; Test type: Other; Effect size (Hedge's g) = 0.36, 95% CI 2-sided [-0.29 to 1.01]
Statistical Analysis 2: Comparison: Intervention; Effect size calculation from Time 1 to Time 3 on P-PRFQ; Test type: Other; Effect size (Hedge's g) = 0.49, 95% CI 2-sided [-0.20 to 1.17]

3. Secondary Outcome: Change on Edinburgh Postnatal Depression Scale (EPDS)
Description: The Edinburgh Postnatal Depression Scale (EPDS; Cox, Holden & Sagovsky, 1987) is a 10-item self-report measure used to identify depression in women during the perinatal period. The scale was initially developed to screen for postnatal depression but has also been validated for use in antenatal populations (Murray & Cox, 1990). Higher total scores indicate higher presence of depressive symptoms i.e. a worse outcome (range 0-30).
Time Frame: Baseline, up to 48-hours post-intervention, 1-month follow-up
Population: N=1 delivered their baby before fully completing Time 2 and therefore did not complete the EPDS at Time 2 or 3. The N=3 who delivered their babies between Time 2 and Time 3 (and therefore did not complete the MAAS and P-PRFQ) still completed the EPDS at Time 3, as it is appropriate to be used in the postnatal period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
score on a scale
  Time 1 (pre-intervention) | 17.3 (3.0)
  Time 2 (up to 48-hours post-intervention): number analyzed (Participants) | 18
  Time 2 (up to 48-hours post-intervention) | 12.1 (4.0)
  Time 3 (1-month follow-up): number analyzed (Participants) | 18
  Time 3 (1-month follow-up) | 10.4 (3.6)
Statistical Analysis 1: Comparison: Intervention; Effect size calculation from Time 1 to Time 2 on EPDS; Test type: Other; Effect size (Hedge's g) = 1.48, 95% CI 2-sided [0.75 to 2.21]
Statistical Analysis 2: Comparison: Intervention; Effect size calculation from Time 1 to Time 3 on EPDS; Test type: Other; Effect size (Hedge's g) = 2.08, 95% CI 2-sided [1.28 to 2.88]

ADVERSE EVENTS:
Time Frame: 4 weeks after attending intervention
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
As this was a small, uncontrolled feasibility study, it is not possible to conclude that any observed changes in prenatal bonding, parental RF or depressive symptomatology were due to the intervention. Future research is needed with larger sample sizes, powered to test for statistically significant changes, and utilising a control condition. A comparison group would allow for greater control of confounding variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT05628675/Prot_SAP_000.pdf